CLINICAL TRIAL: NCT01616303
Title: Phase 2: A Randomized Controlled Study on Effectiveness of Chemotherapy (Carboplatin-Paclitaxel) Versus Chemo-immunotherapy (Carboplatin-Paclitaxel-Oregovomab) in Patients With Advanced Epithelial Ovarian, Adnexal or Peritoneal Carcinoma
Brief Title: A Controlled Study of the Effectiveness of Oregovomab (Antibody) Plus Chemotherapy in Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quest PharmaTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QPT-ORE-002; 2010-024305-13 (EudraCT Number)
Record Dates: First submitted 2012-05-30; First posted 2012-06-11 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Neoplasms
Keywords: ovarian; cancer; neoplasm; adenocarcinoma; CA125
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Adenocarcinoma | interventions — Carboplatin; Paclitaxel; oregovomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- carboplatin & paclitaxel (Active Comparator): first-line chemotherapy for ovarian cancer
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- carboplatin & paclitaxel & oregovomab (Experimental): first-line chemotherapy for ovarian cancer plus oregovomab
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Biological: oregovomab

INTERVENTIONS:
Drug: Carboplatin — carboplatin (area under the curve (AUC) 6, administered intravenously in a single day for 6 cycles every three weeks [21 days])
Drug: Paclitaxel — Paclitaxel (175 mg / square meter, intravenously over three hours in one day to be repeated for 6 cycles every three weeks [21 days])
Biological: oregovomab — oregovomab (2 mg infused intravenously jointly during the 1st, 3rd and 5th chemotherapy cycle and 12 weeks after the 5th cycle).
  Other Names: OvaRex
  Arms: carboplatin & paclitaxel & oregovomab

SUMMARY:
This is a Phase 2 randomized study with two treatment arms to compare the effectiveness of oregovomab (a murine monoclonal antibody directed against cancer antigen 125 (CA125)) when combined with first-line chemotherapy (carboplatin and paclitaxel) to first-line chemotherapy (carboplatin and paclitaxel alone) in female patients with advanced ovarian cancer.

DETAILED DESCRIPTION:
Oregovomab is an investigational drug previously used in clinical trials as an immunotherapeutic treatment of ovarian cancer patients whose tumor cells express the tumor associated antigen, CA125. The active component of oregovomab is the activated murine monoclonal antibody B43.13, an immunoglobulin G1k (IgG1k) subclass immunoglobulin that binds with high affinity (1.16E10/M) to CA125.

CA125 is a surface glycoprotein antigen that is expressed on more than 80% of all non-mucinous epithelial ovarian carcinomas where it occurs at elevated levels in the serum of patients with ovarian cancer. Little is known about its biological function. CA125 is associated with a large molecular weight mucin-like glycoprotein complex of 200-250 kilodaltons (kDa) and its genetic structure has recently been elucidated. There is good evidence to suggest that CA125 is a relevant target antigen for antigen-mediated immunotherapy of ovarian cancer.

The study will compare the effectiveness of oregovomab (a murine monoclonal antibody directed against cancer antigen 125 (CA125)) when combined with first-line chemotherapy (carboplatin and paclitaxel) to first-line chemotherapy (carboplatin and paclitaxel alone) in female patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* have newly diagnosed epithelial adenocarcinoma of ovarian, tubal or peritoneal origin and French Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) Stage III/IV disease.
* have preoperative CA125 levels > 50 U/mL
* have optimal cytoreduction (RT<1)
* be anticipated to have first-line chemotherapy infusion within 6 weeks after surgery
* be available to complete the protocol for the duration of the study
* have adequate Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/µL, equivalent to Common Terminology Criteria (CTCAE v3.0) grade 1. Platelets greater than or equal to 100,000/µL; hemoglobin greater than or equal to 8.0 g/dL
* have adequate Renal function: creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v3.0 grade 1
* have adequate Hepatic function: bilirubin less than or equal to 1.5 x ULN (CTCAE v3.0 grade 1). SGOT and alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* able to sign informed consent and provide authorization permitting release of personal health information
* have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* have an active autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), ankylosing spondylitis)
* have a known allergy to murine proteins or have had a documented anaphylactic reaction to any drug, or cannot tolerate cyclophosphamide
* are being chronically treated with immunosuppressive drugs such as cyclosporin, adrenocorticotropic hormone (ACTH), or systemic corticosteroids.
* have a recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia
* have an acquired, hereditary, or congenital immunodeficiency
* have uncontrolled diseases other than cancer
* have contraindications to the use of pressor agents
* have undergone more than one surgical debulking
* have hepatic dysfunction, eg, bilirubin more than 1.5 times higher than normal levels, lactate dehydrogenase (LDH), serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) doubled compared to normal or albumin <3.5 g/dL
* have severe renal insufficiency with serum creatinine >1.6 mg/dL
* have concomitant diseases or treatments that may confound the results of the study, which may preclude the completion of the protocol or may mask adverse reactions
* are to be tested with other medications during treatment
* are unable to read or understand or unable to sign the necessary written consent before starting treatment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
CA125 ELISPOT assay response for cytotoxic T cell antigen specific immunity induction to end of first-line chemotherapy | At Baseline (up to 4 weeks before Cycle 1), at Cycle 5 (approximately 12 weeks after Cycle 1) and termination (approximately 25 weeks after Cycle 1)
  Change from baseline CA125 ELISPOT assay after stimulation with oregovomab (MAb-B43.13 against CA125) measured at approximately 12 weeks and 25 weeks after the start of first-line chemotherapy

SECONDARY OUTCOMES:
Time to clinical relapse | Up to three years after treatment in the study
  The time period from the date of randomization to the date of confirmed relapse as defined by clinical, radiologic, and/or pathologic evaluations.
Immune parameters: HAMA (human anti-mouse antibody) titers and DTH (delayed type hypersensitivity) | Up to three years after treatment in the study
  Laboratory test for human anti-mouse antibody (HAMA) present in patients' sera. DTH (delayed type hypersensitivity) is an on-site test conducted by the investigator by injecting a small amount of the Oregovomab product and three other antigens (mumps, tetanus, and Candida) into the skin of the patient and observing the effects.
Clinical response | Up to three years after treatment in the study
  Patients will be categorized into one of the following: increasing disease, stable disease, or progression [measurable disease studies]
Overall Survival | Up to three years after treatment in the study
  The observed length of life from entry into the study to death or the date of last contact

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Woo, M.Sc., Study Director — Quest PharmaTech Inc.; Christopher Nicodemus, MD FACP, Study Chair — AIT Strategies
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brewer M, Angioli R, Scambia G, Lorusso D, Terranova C, Panici PB, Raspagliesi F, Scollo P, Plotti F, Ferrandina G, Salutari V, Ricci C, Braly P, Holloway R, Method M, Madiyalakan M, Bayever E, Nicodemus C. Front-line chemo-immunotherapy with carboplatin-paclitaxel using oregovomab indirect immunization in advanced ovarian cancer: A randomized phase II study. Gynecol Oncol. 2020 Mar;156(3):523-529. doi: 10.1016/j.ygyno.2019.12.024. Epub 2020 Jan 6. PMID 31916979
- [Result] Battaglia A, Buzzonetti A, Fossati M, Scambia G, Fattorossi A, Madiyalakan MR, Mahnke YD, Nicodemus C. Translational immune correlates of indirect antibody immunization in a randomized phase II study using scheduled combination therapy with carboplatin/paclitaxel plus oregovomab in ovarian cancer patients. Cancer Immunol Immunother. 2020 Mar;69(3):383-397. doi: 10.1007/s00262-019-02456-z. Epub 2020 Jan 3. PMID 31897661
- See also: Sponsor website — http://www.questpharmatech.com/